CLINICAL TRIAL: NCT02797340
Title: Metformin in Patients With Chronic and Acute Heart Failure: Pharmacokinetics and Polymorphisms in Genes Encoding Membrane Metformin Transporter Proteins
Brief Title: Metformin Pharmacokinetics in Patients With Chronic and Acute Heart Failure
Acronym: MetKin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Wiggers, Senior consultant, associate professor, PhD, DMSc, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 50268-20150921
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — Blood Specimen Collection; Metformin

ARMS (1):
- Interventional (Experimental): All participants
  Interventions: Other: Blood draws and urine samples for metformin concentration measurements; Drug: Metformin

INTERVENTIONS:
Other: Blood draws and urine samples for metformin concentration measurements
Drug: Metformin

SUMMARY:
The study evaluates the pharmacokinetics of metformin in heart failure patients in acute and chronic state in relation to metformin transporter genotypes. Participants have heart failure and type 2 diabetes treated with metformin.

Hypothesis:

Primary: The renal clearance of metformin is decreased in acute state of congestive heart failure compared with chronic state.

Secondary: Metformin trough values in HF patients are influenced by polymorphisms in transporter genes relevant to the pharmacokinetics of metformin.

DETAILED DESCRIPTION:
Background: Heart failure (HF) is a common disease and diabetes/insulin resistance are present in approximately 50 % of HF patients. Metformin is the most commonly prescribed oral anti-diabetic drug, and a huge inter-individual variability in trough steady-state metformin concentration in type 2 diabetics have been demonstrated. Genetic polymorphisms in metformin transporter genes are likely to have a direct impact on metformin pharmacokinetics and variability in drug responses, but the influence of polymorphisms in these transporter genes on circulating metformin levels is presently unknown in HF patients.

Objectives:

A) To compare the pharmacokinetics of metformin in 12 diabetic patients with HF in acute and chronic state.

B) To investigate the influence of polymorphisms in genes encoding the metformin transporter proteins on metformin trough levels in 150 diabetic HF patients.

Design: An open, single-center study enrolling 12 patients with acute heart failure (study A) and 150 patients with stable chronic heart failure (study B). The participants have diabetes already treated with metformin prior to inclusion. Through repeated blood draws, the concentration of metformin will be determined along with genotyping for metformin transporter genes.

Primary outcome:

Study A: Changes in renal clearance of metformin between patients with acute and chronic heart failure.

Study B: Mean trough steady-state concentrations of metformin with emphasis on the intra-interindividual variability in HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure
* LVEF < 45% within 12 months prior to inclusion
* NYHA-class I, II, III or IV
* Ability to understand the written patient information and to give informed consent
* Diabetes Type 2 (and in metformin treatment for > 1 month)
* Stable dosage of metformin treatment for at least 1 week prior to examination

Exclusion Criteria:

* Age < 18 years
* Current abuse of alcohol or drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-01-11 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in renal clearance of metformin between patients with acute and chronic heart failure. | approximately 2 weeks
Mean trough steady-state concentrations of metformin with emphasis on the intra-interindividual variability in HF patients | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark